CLINICAL TRIAL: NCT01141361
Title: Feasibility of Home-based Measurement of Walking Capacity Using Global Positioning System in Patients With Peripheral Arterial Disease
Brief Title: Feasibility of Home-based Measurement of Walking Capacity Using Global Positioning System in Peripheral Artery Disease
Acronym: POST-GPS
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Région des Pays de la Loire (Unknown)
Responsible Party: Sponsor
Other Study IDs: POST-GPS
Record Dates: First submitted 2010-06-08; First posted 2010-06-10 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Peripheral Artery Disease
Keywords: Claudication; Artery; Ambulatory technique; GPS
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Peripheral arterial disease patients: Patients with a peripheral arterial disease, defined by an ankle to brachial index below 0.90
  Interventions: Procedure: GPS recording(s) of walking capacity in PAD patients

INTERVENTIONS:
Procedure: GPS recording(s) of walking capacity in PAD patients — Home-based GPS recording(s) of walking capacity in PAD patients. Two evaluations will be performed. The second evaluation will be performed six months after the initial assessment (test 1) and only for patients with GPS maximal walking distance below 2000 meters at test 1. It is expected that some patients at test 2 will have undergo surgery or endovascular treatment.
  Other Names: Ambulatory technique; Clinical routine

SUMMARY:
The purpose of this study is to assess the feasibility of home-based measurement of walking capacity in peripheral arterial disease (PAD) patients, uing the Global Positioning System (GPS). This study should state if the GPS technique could be used in clinical routine in order to assess walking capacity in PAD patients. Patients will be assessed a first time (test 1) and six months later (test 2).

DETAILED DESCRIPTION:
The measurement of walking capacity in PAD patients is an important step in the management of such patients. The gold standard method to assess this walking capacity is the measurement of the maximal walking distance on a treadmill. However, treadmill measurement are not readily accessible and the relationship with free-living walking capacity is, although not well known, weak. A novel approach was developed using a Global Positioning System in order to assess community-based walking capacity. This method showed interesting results, validating the technique, but was limited to one laboratory and to the place where the measurements were performed. The next step is therefore to assess the feasibility of home-based measurement of walking capacity using the GPS technique, through a multicenter study regrouping university hospitals, independent vascular specialists (angiologists) and private clinic(s).

ELIGIBILITY:
Inclusion Criteria:

* ABI < 0.90 or patients with vascular history (surgery, endovascular treatment) and having vascular type claudication
* Older than 18 years
* Vascular-type claudication (defined by the Leriche classification and the Edimbourg questionnaire criterion)
* Informed consent of the patient

Non-Inclusion Criteria:

* No informed consent of the patient
* Exercise (walking) limitation other than vascular explained limitation
* Critical limb ischemia (Leriche stage 3 or 4)
* Major cardiovascular events in the last 3 months
* Pregnant woman
* Patient unable to understand the protocol of the study

Exclusion Criteria:

* Withdrawal of the informed consent of the patient following the inclusion period
* Emergence of a non-inclusion criteria during the inclusion period
* Patient with a GPS maximal walking distance > 2000 meters following the first evaluation (can not be considered as having a major walking limitation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral arterial disease, defined by an ankle to brachial index below 0.90, or patients with vascular history and having vascular claudication
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2009-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Percentage of home-based GPS recordings that are analyzable | December 2011

SECONDARY OUTCOMES:
"Technical quality" of recorded GPS signals | December 2011
Easiness of the interpretation of the GPS measurements | December 2011
Adherence of the patients to the protocol | December 2011
Compare GPS results to the results obtained with different questionnaires (external validity) | December 2011
  The questionnaires used assess the physical activity level, the quality of life and the walking impairment of the studied PAD patients.
Sensibility of GPS measurements after (or not) a therapeutic treatment (endovascular treatment, surgery) | December 2011

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Abraham, MD, PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- University Hospital, Angers, France

REFERENCES:
- [Derived] Gernigon M, Le Faucheur A, Fradin D, Noury-Desvaux B, Landron C, Mahe G, Abraham P. Global positioning system use in the community to evaluate improvements in walking after revascularization: a prospective multicenter study with 6-month follow-up in patients with peripheral arterial disease. Medicine (Baltimore). 2015 May;94(18):e838. doi: 10.1097/MD.0000000000000838. PMID 25950694